CLINICAL TRIAL: NCT03037099
Title: Enhancing Glycemic Index Knowledge and Application Among Adults With Type-2 Diabetes Mellitus
Brief Title: Healthy Eating and Active Living for Diabetes: Glycemic Index
Acronym: HEALD-GI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Athabasca University (Other)
Collaborators: University of Alberta (Other); Canadian Foundation for Dietetic Research (CFDR) (Other)
Responsible Party: Principal Investigator, Steven T. Johnson, Associate Professor, Athabasca University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HEALD-GI
Record Dates: First submitted 2016-08-18; First posted 2017-01-31 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes
Keywords: Glycemic index; dietary intakes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced GI Concept Education (Experimental): This group will receive enhanced GI concept nutrition education including GI values of foods, low GI recipes, menus, and application through websites with chat rooms, online videos and print materials. These will be reinforced through email, text messaging/phone calls, and postal mail.
  Interventions: Behavioral: Enhanced GI Concept Education
- Usual Care (No Intervention): Usual care group will receive only standard printed copies of Canada Food Guide and Canadian Diabetes Association GI resources.

INTERVENTIONS:
Behavioral: Enhanced GI Concept Education
  Arms: Enhanced GI Concept Education

SUMMARY:
The main purpose of this study is to examine the effectiveness of enhanced GI-targeted nutrition education on dietary behaviour and intakes among adults with type 2 diabetes. Sixty-six eligible participants will be randomized into two equal groups using a pragmatic randomized controlled trial design.

DETAILED DESCRIPTION:
This study proposes to examine the effectiveness of enhanced GI-targeted nutrition education on dietary behaviour and intakes among adults with type 2 diabetes.

Adults with type 2 diabetes will take part in this study and will be randomly assigned to either the HEALD-GI program (intervention) or in usual care (control). To evaluate the effectiveness of the program, 66 eligible participants drawn from the Alberta's Caring for Diabetes Cohort will be randomized into two equal groups using a pragmatic randomized controlled trial design. The control will receive only standard printed copies of Canada Food Guide and Canadian Diabetes Association (CDA) GI resources. The intervention group will receive additional GI concept information including GI values of foods, low GI recipes, menus, and application through websites with chat rooms, online videos, and print materials. These will be reinforced through email, text messaging/phone calls, and postal mail. GI knowledge and skill, self-efficacy, dietary intakes (using 3-day food record), anthropometry (body mass), and clinical measures (glycated hemoglobin A1c, systolic blood pressure), will be assessed at baseline and three months post-intervention.

The primary outcome will be change in GI related dietary behaviour and intake measured using 3-day food records (baseline and 3 months). Secondary outcomes include: 1) body mass, 2) glycemic control (hemoglobin A1c), 3) systolic blood pressure.

Significance:

Sufficient evidence is needed regarding the best approach for increasing uptake of current Canadian Diabetes Association (CDA) evidence-based recommendation to include low GI foods in daily meal planning as an effective dietary self-care practice for glycemic control among people with type 2 diabetes. Findings from this study will help determine if, and how, the current approach to disseminating the CDA dietary recommendations pertaining to GI concept could be improved for better uptake using the most efficient and cost effective patient-centered approaches to nutrition self-management. Besides, evidence generated will contribute to addressing some of the controversies regarding the clinical usefulness of the GI concept.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 years of age or older; identified as having T2DM and currently enrolled in the Alberta's Caring for Diabetes cohort study
* Able to read, understand, and converse in English
* Willing to provide informed consent and currently living in Edmonton.

Exclusion Criteria:

* Those taking exogenous insulin and having physiological and /or medical conditions that interfere with normal digestive functions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Dietary glycemic index | 12 weeks
  arbitrary units

SECONDARY OUTCOMES:
Body mass | 12 weeks
  kilograms
Glycemic control (hemoglobin A1c) | 12 weeks
Systolic blood pressure | 12 weeks
  mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Steven T Johnson, PhD, Principal Investigator — Athabasca University
Locations (2):
- Canada (2):
  - Athabasca University, Athabasca, Alberta
  - Alliance for Canadain Health Outcomes Research in Diabetes, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al Sayah F, Majumdar SR, Soprovich A, Wozniak L, Johnson ST, Qiu W, Rees S, Johnson JA. The Alberta's Caring for Diabetes (ABCD) Study: Rationale, Design and Baseline Characteristics of a Prospective Cohort of Adults with Type 2 Diabetes. Can J Diabetes. 2015 Oct;39 Suppl 3:S113-9. doi: 10.1016/j.jcjd.2015.05.005. Epub 2015 Aug 1. PMID 26243463
- See also: Research group — http://www.achord.ca